CLINICAL TRIAL: NCT03377647
Title: An Asthma Collaboration to Reduce Childhood Asthma Disparities on the Navajo Nation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HS2970
Record Dates: First submitted 2017-11-01; First posted 2017-12-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Year two intervention (Active Comparator): Both interventions will occur in the Tuba City Agency during year two.
  Interventions: Behavioral: Asthma Care Provider Training; Behavioral: School Staff Asthma Education
- Year three intervention (Active Comparator): Both interventions will occur in the Chinle Agency during year three.
  Interventions: Behavioral: Asthma Care Provider Training; Behavioral: School Staff Asthma Education
- Year four intervention (Active Comparator): Both interventions will occur in the Fort Defiance during year four.
  Interventions: Behavioral: Asthma Care Provider Training; Behavioral: School Staff Asthma Education

INTERVENTIONS:
Behavioral: Asthma Care Provider Training — In this intervention, asthma care providers will be trained in current, evidence-based guidelines for care of children with asthma, and will be provided with tools that their practice may use to facilitate care improvements.
Behavioral: School Staff Asthma Education — In this intervention, teachers and other school staff will be provided current, evidence-based training in understanding asthma and will be provided tools to help schools address the special needs of children with asthma.

SUMMARY:
National Jewish Health and The University of Arizona worked with Navajo Nation organizations to develop this program to improve the health of children with asthma. The Navajo Community Asthma Program will have two main parts. One will train doctors and health care professionals to improve the diagnosis and treatment of asthma. The second part will work with area schools to provide education to school nurses, teachers, and children to help them better understand asthma. The project also works with families to help them know how to best take care of their child's asthma. A major project aim is to make sure that doctors, teachers, and families work together to manage asthma.

ELIGIBILITY:
The project will involve three Navajo Nation Agencies: Tuba City, Chinle, and Fort Defiance. Project interventions will run for one year in each Agency. Interventions are population-level interventions. No intervention will be administered at the individual level.

Inclusion Criteria:

- The study will be conducted within three agencies on the Navajo Nation, each of which has its own IHS service unit. The three agencies are Chinle, Tuba City, and Fort Defiance.

Exclusion Criteria:

- This protocol pertains only to the three agencies listed above.

Community interviewees will be interested candidates who meet the following eligibility criteria:

Inclusion Criteria:

1. Able and willing to provide informed consent
2. Greater than or equal to 18 years of age
3. Guardianship of a child younger than 18 years of age who has been diagnosed with asthma
4. Able to read and/or understand English or Navajo

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Younger than 18 years of age, without presence of guardian
3. Unable to read and/or understand English or Navajo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of pediatric asthma exacerbations in Year 1 | Data will be collected once during Year 1 of the project.
  The rate of asthma exacerbations among children living on the Navajo Nation during Year 1 of the project as measured by hospitalizations and urgent care visits. This rate will be assessed by review of Indian Health Service (IHS) data.
Rate of pediatric asthma exacerbations in Year 2 | Data will be collected once during Year 2 of the project.
  The rate of asthma exacerbations among children living on the Navajo Nation during Year 2 of the project as measured by hospitalizations and urgent care visits. This rate will be assessed by review of Indian Health Service (IHS) data.
Rate of pediatric asthma exacerbations in Year 3 | Data will be collected once during Year 3 of the project.
  The rate of asthma exacerbations among children living on the Navajo Nation during Year 3 of the project as measured by hospitalizations and urgent care visits. This rate will be assessed by review of Indian Health Service (IHS) data.
Rate of pediatric asthma exacerbation in Year 4 | Data will be collected once during Year 4 of the project.
  The rate of asthma exacerbations among children living on the Navajo Nation during Year 4 of the project as measured by hospitalizations and urgent care visits. This rate will be assessed by review of Indian Health Service (IHS) data.
Rate of pediatric asthma exacerbations in Year 5 | Data will be collected once during Year 5 of the project.
  The rate of asthma exacerbations among children living on the Navajo Nation during Year 5 of the project as measured by hospitalizations and urgent care visits. This rate will be assessed by review of Indian Health Service (IHS) data.
Rate of pediatric asthma exacerbations in Year 6 | Data will be collected once during Year 6 of the project.
  The rate of asthma exacerbations among children living on the Navajo Nation during Year 6 of the project as measured by hospitalizations and urgent care visits. This rate will be assessed by review of Indian Health Service (IHS) data.

SECONDARY OUTCOMES:
Community reports of asthma-related events Year 1 | In-person interviews will be conducted with families during year one of the project.
  Families will be interviewed to assess child asthma symptom control and related care satisfaction.
Community reports of asthma-related events Year 2 | In-person interviews will be conducted with families during year two of the project.
  Families will be interviewed to assess child asthma symptom control and related care satisfaction.
Community reports of asthma-related events Year 3 | In-person interviews will be conducted with families during year three of the project.
  Families will be interviewed to assess child asthma symptom control and related care satisfaction.
Community reports of asthma-related events Year 4 | In-person interviews will be conducted with families during year four of the project.
  Families will be interviewed to assess child asthma symptom control and related care satisfaction.
Community reports of asthma-related events Year 5 | In-person interviews will be conducted with families during year five of the project.
  Families will be interviewed to assess child asthma symptom control and related care satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bender, PhD, Principal Investigator — National Jewish Health
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - National Jewish Health, Denver, Colorado

REFERENCES:
- [Derived] Lowe AA, Ravi P, Hudson B, Begay E, Tso B, Liu AH, Bender BG, Gerald LB, King DK. Using document analysis methods and implementation science frameworks to conduct a process evaluation of the community asthma program on the Navajo Nation. Transl Behav Med. 2025 Jan 16;15(1):ibaf056. doi: 10.1093/tbm/ibaf056. PMID 41027683